CLINICAL TRIAL: NCT00635765
Title: Open Label Extension Study Evaluating the Safety and Biological Activity of a New Prolonged Release Formulation of Octreotide Acetate, C2L-OCT-01 PR, Administered Intra Muscularly Every 6, 5 or 4 Weeks in Acromegalic Patients
Brief Title: Open Label Extension Study Evaluating Safety and Biological Activity of C2L-OCT-01 PR in Acromegalic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ambrilia Biopharma, Inc. (Industry)
Responsible Party: Bonabes de Rouge, M.D./Senior Executive Vice-President & Chief Scientist Officer, Ambrilia Biopharma, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2L-OCT-01 PR-302
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: C2L-OCT-01 PR 30 mg — Administered by deep IM (gluteus) on Day 1. Beginning on Day 42, drug injection frequency (6, 5 or 4 weeks) and dose modification/adjustment will be allowed for every 3 drug injections based on the mean serum GH and clinical symptoms obtained at the last visit of study C2L-OCT-01 PR-301 and during the course of this study.

SUMMARY:
The purpose of this study is to assess the safety profile of C2L-OCT-01 PR for up to an additional 96-week period in acromegalic patients who completed the C2L-OCT-01 PR-301 study.

ELIGIBILITY:
Inclusion Criteria:

•Subjects who have completed the 24-week C2L-OCT-01 PR-301 study

Exclusion Criteria:

* Women of childbearing potential who are not taking adequate contraception or who are pregnant or lactating
* Subjects who have experienced any clinically significant adverse event related to study medication in C2L-OCT-01 PR-301 study
* Subjects with uncontrolled Diabetes type II
* Subjects with signs or symptoms related to a tumor compression of the optical chiasm
* Subjects with symptomatic cholelithiasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Assess, for up to an additional 96 weeks, the safety profile of C2L-OCT-01 PR administered intra muscularly every 6, 5 or 4 weeks in patients who have completed the C2L-OCT-01 PR-301 study. | Up to 96 weeks

SECONDARY OUTCOMES:
To determine the percentage of patients who remain with controlled mean GH and normal (gender- and age-matched values) IGF-1 serum concentrations. | Up to 96 weeks
Compare plasma concentrations of C2L-OCT-01 PR. | First 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Naudin, M.D., Study Director — Ambrilia Biopharma, Inc.
Locations (6):
- Republican Centre for Medical Rehabilitation and Water-therapy, Minsk, Belarus
- Semmelweis Egyetem Altalanos Orvostudomanyi, Budapest, Hungary
- Institue of Endocrinology "C.I Parhon" Bucharest, Bucharest, Romania
- Institute of Endocrinology, University Clinical Center, Belgrade, Serbia
- Fakultna Nemocnica s Poliklinkow Bratislava, Bratislava, Slovakia
- V.P. Komisarenko Institute of Endocrinology and Metabolism, AMS Ukraine, Kiev, Ukraine